CLINICAL TRIAL: NCT00317811
Title: A Phase II Trial of Bortezomib + Ascorbic Acid + Melphalan (BAM) Combination Therapy for Patients With Newly Diagnosed Multiple Myeloma
Brief Title: Bortezomib, Ascorbic Acid, and Melphalan in Treating Patients With Newly Diagnosed Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oncotherapeutics (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000479708; ONCOTHER-20052183; ONCOTHER-BAM2005; MILLENNIUM-ONCOTHER-20052183
Record Dates: First submitted 2006-04-24; First posted 2006-04-25 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2011-06

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Ascorbic Acid; Bortezomib; Melphalan

INTERVENTIONS:
Dietary Supplement: ascorbic acid
Drug: bortezomib
Drug: melphalan

SUMMARY:
RATIONALE: Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as melphalan, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Ascorbic acid may help melphalan work better by making cancer cells more sensitive to the drug. Giving bortezomib together with ascorbic acid and melphalan may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving bortezomib together with ascorbic acid and melphalan works in treating patients with newly diagnosed multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the overall response rate (combined complete response [CR], near CR, partial response [PR], and minimal response [MR]) and time to progression of disease in patients with newly diagnosed multiple myeloma treated with bortezomib, ascorbic acid, and melphalan.
* Assess the safety and tolerability of this regimen in these patients.

Secondary

* Assess the time to response in these patients.
* Determine progression-free and overall survival of these patients.
* Assess time to disease progression among subjects who continue to maintenance treatment with bortezomib.

OUTLINE: This is an open-label study.

* Induction therapy: Patients receive bortezomib IV on days 1, 4, 8, and 11 and oral melphalan and oral ascorbic acid on days 1-4. Treatment repeats every 28 days to maximum response [MR] or for at least 8 courses in the absence of disease progression or unacceptable toxicity. Patients with responding disease receive an additional 2 courses of induction therapy beyond MR and proceed to maintenance therapy. Patients with stable disease or without a maximum reduction in their paraprotein after 8 courses of induction therapy are eligible to receive maintenance therapy.
* Maintenance therapy: Patients receive bortezomib IV on days 1 and 15. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 35 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed symptomatic multiple myeloma based on the following criteria:

  * Durie-Salmon staging
  * Measurable disease, defined as a monoclonal immunoglobulin spike on serum electrophoresis of ≥ 1 g/dL and/or urine monoclonal immunoglobulin spike of ≥ 200 mg/24 hours
* Symptomatic disease
* No POEMS syndrome (plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein [M-protein], and skin changes)
* No plasma cell leukemia

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* Life expectancy > 3 months
* Platelet count ≥ 50,000/mm³ (30,000/mm³ if the bone marrow is extensively infiltrated)
* Hemoglobin ≥ 8.0 g/dL
* Absolute neutrophil count ≥ 1,000/mm³
* Creatinine ≤ 3 mg/dL
* Sodium > 130 mmol/L corrected
* AST and ALT ≤ 3 times upper limit of normal (ULN)
* Bilirubin ≤ 2 times ULN unless clearly related to the disease
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Any ECG abnormality has to be documented by the investigator as not medically relevant
* No electrocardiographic evidence of acute ischemia or new conduction system abnormalities
* No myocardial infarction or EKG evidence of infarction within the past 6 months
* No active infection
* No severe hypercalcemia (i.e., serum calcium ≥ 14 mg/dL [3.5 mmol/L])
* No New York Heart Association class III or IV heart failure
* No uncontrolled angina
* No severe uncontrolled ventricular arrhythmias
* No active conduction system abnormalities
* No poorly controlled hypertension
* No diabetes mellitus
* No known HIV infection
* No known active hepatitis B or C viral infection
* No history of grand mal seizures
* No history of allergic reaction to compounds of similar chemical or biological composition to melphalan, bortezomib, boron, or mannitol
* No peripheral neuropathy ≥ grade 2 within the past 14 days
* No other serious medical or psychiatric illness that could potentially interfere with the completion of study treatment

PRIOR CONCURRENT THERAPY:

* More than 4 weeks since prior immunotherapy, antibody therapy, or radiotherapy
* More than 4 weeks since prior major surgery
* No prior therapy for myeloma

  * Prior prednisone at a total of 400mg over ≤ 4 days (or an equivalent potency of another steroid) allowed
* No concurrent corticosteroids (≥ 10 mg prednisone/day or equivalent)
* No other concurrent investigational agents
* No other concurrent antimyeloma therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2005-11; Primary Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Overall response rate (complete response [CR], near CR, partial response, and minimal response)
Safety and tolerability as assessed by NCI CTCAE v3.0
Proportion of patients responding
Time to disease progressionin patients receiving maintenance treatment

SECONDARY OUTCOMES:
Time to response
Progression-free survival
Overall survival as assessed by the Kaplan-Meier method
Time to disease progression

CONTACTS AND LOCATIONS:
Overall Officials: James R. Berenson, MD, Principal Investigator — Oncotherapeutics
Locations (8):
- United States (8):
  - Hematology-Oncology Medical Group of Fresno, Incorporated, Fresno, California
  - Hematology Oncology Medical Group of Orange County, Incorporated, Orange, California
  - Oncotherapeutics, West Hollywood, California
  - Florida Cancer Specialists - Bonita Springs, Bonita Springs, Florida
  - Florida Oncology Associates, Orange Park, Florida
  - Atlanta Cancer Care - Roswell, Roswell, Georgia
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - SUNY Downstate Medical Center, Brooklyn, New York

REFERENCES:
- [Result] Berenson JR, Yellin O, Woytowitz D, Flam MS, Cartmell A, Patel R, Duvivier H, Nassir Y, Eades B, Abaya CD, Hilger J, Swift RA. Bortezomib, ascorbic acid and melphalan (BAM) therapy for patients with newly diagnosed multiple myeloma: an effective and well-tolerated frontline regimen. Eur J Haematol. 2009 Jun;82(6):433-9. doi: 10.1111/j.1600-0609.2009.01244.x. Epub 2009 Feb 17. PMID 19226361